CLINICAL TRIAL: NCT03755037
Title: Clomiphine Citrate and Estradiol Versus Clomiphine Citrate and Sildenafil in Comparison With Clomiphine Citrate Alone for Induction of Ovulation in Unexplained Infertility: Double Blind Randomised Trial
Brief Title: Clomiphene Citrate, Estradiol and Sildenafil for Induction of Ovulation in Unexplained Infertility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nesreen Abdel Fattah Abdullah Shehata (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Sponsor-Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assistant professor, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Beni-Suef 16
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Clomiphene; Ethinyl Estradiol

STUDY DESIGN:
Intervention Model Description: Women with unexplained infertility (n=150) were divided into 3 equal groups. Group 1 received estradiol and clomiphine citrate (cc), group 2 received sildenafil and cc and group 3 cc and placebo.
Who Masked: Participant, Investigator
Masking Description: Double blind randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Estradiol and cc (Active Comparator): Group 1 received estradiol, cc and placebo simillar to sildenafil for induction of ovulation.
  CC 50 mg (clomid) orally twice daily from 3rd day to 7th day of menstrual cycle of the patient then ethinyl estradiol 0.05mg orally twice daily on the 8th day of same cycle till 11th day.
  Interventions: Drug: Clomid, Respatio and Ethinyl estradiol
- Sildenafil and cc (Active Comparator): Group 2 received CC 50 mg (clomid) orally twice daily from 3rd day to 7th day of menstrual cycle of the patient, sildenafil citrate (Respatio) 20 mg tab orally 3 times daily from8th day of same cycle till 11th day and placebo simillar to estradiol.
  Interventions: Drug: Clomid, Respatio and Ethinyl estradiol
- Placebo and cc (Placebo Comparator): Group 3 received cc and placebo similar to sildenafil and placebo similar to estradiol with the same doses.
  Interventions: Drug: Clomid, Respatio and Ethinyl estradiol

INTERVENTIONS:
Drug: Clomid, Respatio and Ethinyl estradiol — Drugs were received during the menstrual cycle.

SUMMARY:
Diagnosis of unexplained infertility is made after the recommended testing fails to reveal any abnormality. The treatment for unexplained infertility is empiric because it does not address a specific defect or functional impairment. The principal treatments for unexplained infertility include expectant observation with timed intercourse and lifestyle changes, clomiphene citrate and intrauterine insemination (IUI), controlled ovarian hyperstimulation (COH) with IUI, and IVF).

DETAILED DESCRIPTION:
Clomiphene citrate has been widely used alone, and in combination with intrauterine insemination (IUI), for treatment of unexplained subfertility, The mechanism of action is based on its mixed estrogenic and antiestrogenic properties. Clomiphene is frequently used to treat unexplained female infertility by inducing multifollicular response and correcting potential subtle ovulatory dysfunction .,)The American Society for Reproductive Medicine,2003).

The use of clomiphene citrate decreases the uterine blood flow during the early luteal phase, a periimplantation stage., )The American College of Obstetricians and Gynecologists,1995).

Although ovulation is found in 80% of women with a cumulative effect in 6-8 months, the pregnancy rate can still be very low in these women . The possible causes are the anti-estrogenic effects of CC at the endometrium and cervical mucus level . The endometrial effect is without doubt one of the most important handicaps in infertility treatment. The pregnancy rate can be very low, especially if the endometrial thickness (ET) is <6-8 mm ., )J Turk Ger Gynecol Assoc. ,2012).

Ethinyl E2 reverse the deleterious effect of CC on endometrial development during the follicular phase. Endometrial thickness was dependent on peak E2 concentrations in serum.,(Richard P. Dickey, et.al.,2003).

Sildenafil citrate could lead to an improvement in uterine blood flow and, in conjunction with estrogen, led to the estrogen-induced proliferation of the endometrial lining .

Sildenafil citrate enhances uterine blood flow and increases endometrial thickening . The achieved implantation depends on the blastocyst's ability to infiltrate the endometrium and develop a sustaining blood supply, which requires the following genes to produce the necessary proteins for digesting the endometrial cellular matrix, to regulate cell growth, and to induce angiogenesis (Razieh Dehghani Firouzabadi,et.al.,2013).

ELIGIBILITY:
Inclusion Criteria:

* Women whose infertility tests were normal then diagnosed as unexplained infertility.

Exclusion Criteria:

* Any cause of infertility male factor, tubal or ovarian.
* Chronic illness as cardiac or renal disease
* Any contraindication for used drugs

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female unexplained infertility patients
Enrollment: 150 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Ultrasound parameters | at day 14 until day 17 of menstrual cycle
  Number of follicles in each ovary and endometrial thickness

SECONDARY OUTCOMES:
Pregnancy | at day 21 and 24 of menstrual cycle
  A serum pregnancy test was done

CONTACTS AND LOCATIONS:
Locations (1):
- Nesreen Abd El Fattah Abd Allah, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Alexander Quaas, MD, Ph .D .,and Anuja Dokras, MD . diagnosis and treatment of unexplainrd infertilityRev Obstet Gynecol. 2008 Spring; 1(2): 69-76 2. J Turk Ger Gynecol Assoc.: The effect of administering estrogen to clomiphene citrate stimulated cycles on endometrial thickness and pregnancy rates in unexplained infertility. (2012) . Sep 1;13(3):157-61. 3. Paulus WE, Strehler E, Zhang M, Jelinkova L,El-Danasouri I and Sterzik K. : Benefit of sildenafil citrate in assisted reproductivetherapy. Fertil Steri 2002 Apr;77(4):846-7. 4. Razieh Dehghani Firouzabadi, M.D., Robab Davar, M.D., Farzaneh Hojjat, M.D., and Mohamad Mahdavi, M.D. :effect of sildenafil on endomeerial preparation and outcome of frozen_thawed embryo transfer cycles(. Iran J Reprod Med. 2013 Feb; 11(2): 151-158. 5. Richard P. Dickey, M.D., Ph.D.,):clomiphene citrate for woman with unexplained infertility . pp 261-271 13 May 2015 6. The American Society for Reproductive Medicine. Use of clomiphene citrate in infertile women:. Fertil Steril . Fertil Steril. 2013 Aug;100(2):341-8. doi: 10.1016/j.fertnstert.2013.05.033. Epub 2013 Jun 27.